CLINICAL TRIAL: NCT03545295
Title: Determination Of The Relationship Between Local Anesthetic Volume And Its Dispersion In Ultrasound Guided Quadratus Lumborum Block In Cadavers
Brief Title: Determination Of Dispersion In Ultrasound Guided Quadratus Lumborum Block In Cadavers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Marcelo Vaz Perez, Médico Assistente, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Quadratus Lumborum Block
Record Dates: First submitted 2018-05-12; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Nerve Block

STUDY DESIGN:
Intervention Model Description: the cadavers will be randomized to receive the intervention (Quadratus Lumborum Block) by different techniques (QLB 2/ QLB3) and different volumes (10, 20, 30 ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- QLB 2 10ml (Experimental): The cadaver will receive an ultrasound- guided Quadratus Lumborum Block type 2 with 10 ml coloring solution
  Interventions: Procedure: Quadratus Lumborum Block type 2
- QLB 2 20ml (Experimental): The cadaver will receive an ultrasound- guided Quadratus Lumborum Block type 2 with 20 ml coloring solution
  Interventions: Procedure: Quadratus Lumborum Block type 2
- QLB 2 30ml (Experimental): The cadaver will receive an ultrasound- guided Quadratus Lumborum Block type 2 with 30 ml coloring solution
  Interventions: Procedure: Quadratus Lumborum Block type 2
- QLB 3 10ml (Experimental): The cadaver will receive an ultrasound- guided Quadratus Lumborum Block type 3 with 10 ml coloring solution
  Interventions: Procedure: Quadratus Lumborum Block type 3
- QLB 3 20ml (Experimental): The cadaver will receive an ultrasound- guided Quadratus Lumborum Block type 3 with 20 ml coloring solution
  Interventions: Procedure: Quadratus Lumborum Block type 3
- QLB 3 30ml (Experimental): The cadaver will receive an ultrasound- guided Quadratus Lumborum Block type 3 with 30 ml coloring solution
  Interventions: Procedure: Quadratus Lumborum Block type 3

INTERVENTIONS:
Procedure: Quadratus Lumborum Block type 2 — Ultrasound guided injection of coloring solution using a 18g Tuohy echogenic needle, posterior to the Quadratus Lumborum muscle
  Arms: QLB 2 10ml; QLB 2 20ml; QLB 2 30ml
Procedure: Quadratus Lumborum Block type 3 — Ultrasound guided injection of coloring solution using a 18g Tuohy echogenic needle, anterior to the Quadratus Lumborum muscle
  Arms: QLB 3 10ml; QLB 3 20ml; QLB 3 30ml

SUMMARY:
Lumbar Quadrant Blockade is a recent analgesic technique consisting of the injection of local anesthetic around the lumbar square muscle. It was initially described as a technique for abdominal wall analgesia, but later studies have increased the range of indications for laparoscopic and lower limb surgeries. There are several techniques described but with differences in the literature at the point of injection and volume of anesthetic. The exact mechanism of visceral analgesia has not yet been determined. The objective of this study is to determine the dispersion of local anesthetic as a variable dependent on the volume of local anesthetic and injection site and elucidate the mechanisms of analgesia.

DETAILED DESCRIPTION:
After the free and informed consent signed by the family authorizing the procedure, demographic and clinical data will be collected from the medical records of the deceased. The corpse will be weighed, measured and placed on the autopsy table. Blockade randomization (QLB 2 or QLB 3) and volume of local anesthetic (10ml, 20ml, 30ml) will be performed for each side. Injection in the anterior or posterior plane to the Lumbar Quadrant muscle will be performed by anesthesiologists experienced in the technique with ultrasound aid. A colouring solution will be used. After confirming the correct needle position, the previously randomized volumes will be injected. After the blockage, the corpse will be placed in the supine position and will be submitted to autopsy by standard procedure. After removal of the thoracic and abdominal viscera, the investigators will verify the dispersion of the local anesthetic. Photographic records will be made and the number of levels by which the solution dispersed will be annotated, calculating the number of cranial and caudal levels. The corpse will then have its autopsy procedure completed, with the placement of the viscera and incision closure according to the service standard.

ELIGIBILITY:
Inclusion Criteria:

* Fresh corpses - not subjected to a formaldehyde process or frozen for more than 24 hours
* Age ≥ 18 years.
* Free, informed and informed consent signed by relatives or guardians of the body.
* Height> 150 cm and <190 cm

Exclusion Criteria:

* Previous spinal surgery.
* Significant spinal deformity
* Body mass index (BMI) ≥ 35 kg / m2
* Absence of relatives or guardians who can sign the written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Spread of coloring solution according to the volume injected | 3 hours
  Observation of coloring solution around the spinal nerves as they exit the vertebral foramen. Comparison of number of spinal nerves colored according to the volume injected.

SECONDARY OUTCOMES:
Spread of coloring solution to the paravertebral space | 3 hours
  Observation of coloring solution on the paravertebral space. Comparison of spread to the paravertebral space according to the volume injected.
Comparison of spread of the coloring solution between QLB 2 and QLB3 | 3 hours
  Observation of coloring solution around the spinal nerves as they exit the vertebral foramen and spread to the paravertebral space. Comparison of number of spinal nerves colored according to the technique used.

CONTACTS AND LOCATIONS:
Overall Officials: Marilia Tassinari Gonçalves Preza, MD, Principal Investigator — Post Graduate
Locations (1):
- Irmandade de Misericórdia da Santa Casa De São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The research results will be published in indexed scientific journals, maintaining participants identity confidential

REFERENCES:
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] Murouchi T, Iwasaki S, Yamakage M. Quadratus Lumborum Block: Analgesic Effects and Chronological Ropivacaine Concentrations After Laparoscopic Surgery. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):146-50. doi: 10.1097/AAP.0000000000000349. PMID 26735154
- [Background] Tamura T, Kitamura K, Yokota S, Ito S, Shibata Y, Nishiwaki K. Spread of Quadratus Lumborum Block to the Paravertebral Space Via Intramuscular Injection: A Volunteer Study. Reg Anesth Pain Med. 2018 May;43(4):372-377. doi: 10.1097/AAP.0000000000000735. PMID 29389680
- [Background] Wahal C, Kumar A, Pyati S. Advances in regional anaesthesia: A review of current practice, newer techniques and outcomes. Indian J Anaesth. 2018 Feb;62(2):94-102. doi: 10.4103/ija.IJA_433_17. PMID 29491513
- [Background] Elsharkawy H, El-Boghdadly K, Kolli S, Esa WAS, DeGrande S, Soliman LM, Drake RL. Injectate spread following anterior sub-costal and posterior approaches to the quadratus lumborum block: A comparative cadaveric study. Eur J Anaesthesiol. 2017 Sep;34(9):587-595. doi: 10.1097/EJA.0000000000000680. PMID 28731927
- [Background] Dam M, Moriggl B, Hansen CK, Hoermann R, Bendtsen TF, Borglum J. The Pathway of Injectate Spread With the Transmuscular Quadratus Lumborum Block: A Cadaver Study. Anesth Analg. 2017 Jul;125(1):303-312. doi: 10.1213/ANE.0000000000001922. PMID 28277325
- [Background] Hernandez MA, Vecchione T, Boretsky K. Dermatomal spread following posterior transversus abdominis plane block in pediatric patients: our initial experience. Paediatr Anaesth. 2017 Mar;27(3):300-304. doi: 10.1111/pan.13034. Epub 2017 Jan 18. PMID 28098413
- [Background] Oksuz G, Bilal B, Gurkan Y, Urfalioglu A, Arslan M, Gisi G, Oksuz H. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Children Undergoing Low Abdominal Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):674-679. doi: 10.1097/AAP.0000000000000645. PMID 28759502
- [Background] Ishio J, Komasawa N, Kido H, Minami T. Evaluation of ultrasound-guided posterior quadratus lumborum block for postoperative analgesia after laparoscopic gynecologic surgery. J Clin Anesth. 2017 Sep;41:1-4. doi: 10.1016/j.jclinane.2017.05.015. Epub 2017 Jun 1. PMID 28802593
- [Background] Ueshima H, Otake H. RETRACTED: Clinical experiences of unilateral anterior sub-costal quadratus lumborum block for a nephrectomy. J Clin Anesth. 2018 Feb;44:120. doi: 10.1016/j.jclinane.2017.11.031. Epub 2017 Nov 29. No abstract available. PMID 29195100 (Retraction: PMID 35393174 J Clin Anesth. 2022 Aug;79:110749)
- [Background] Ueshima H, Hiroshi O. RETRACTED: Lumbar vertebra surgery performed with a bilateral posterior quadratus lumborum block. J Clin Anesth. 2017 Sep;41:61. doi: 10.1016/j.jclinane.2017.06.012. Epub 2017 Jul 3. No abstract available. PMID 28802611 (Retraction: PMID 35396108 J Clin Anesth. 2022 Aug;79:110790)
- [Background] Ben-David B, La Colla L. Extravasated Fluid in Hip Arthroscopy and Pain: Is Quadratus Lumborum Block the Answer? Anesth Analg. 2017 Jul;125(1):364. doi: 10.1213/ANE.0000000000002198. No abstract available. PMID 28609336
- [Background] Gehling M, Tryba M. Risks and side-effects of intrathecal morphine combined with spinal anaesthesia: a meta-analysis. Anaesthesia. 2009 Jun;64(6):643-51. doi: 10.1111/j.1365-2044.2008.05817.x. PMID 19462494
- [Background] Jeng CL, Torrillo TM, Rosenblatt MA. Complications of peripheral nerve blocks. Br J Anaesth. 2010 Dec;105 Suppl 1:i97-107. doi: 10.1093/bja/aeq273. PMID 21148659
- [Background] Ueshima H, Otake H. RETRACTED: Lower limb amputations performed with anterior quadratus lumborum block and sciatic nerve block. J Clin Anesth. 2017 Feb;37:145. doi: 10.1016/j.jclinane.2016.12.026. Epub 2017 Jan 10. No abstract available. PMID 28235508 (Retraction: PMID 35393170 J Clin Anesth. 2022 Aug;79:110743)